CLINICAL TRIAL: NCT06153979
Title: Investigation of Immune Amnesia Following Measles Infection in Select African Regions
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: Measles West Africa 01
Record Dates: First submitted 2023-10-25; First posted 2023-12-01 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Measles Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and upper respiratory specimens will be stored for analysis in repositories in each participating country.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1 - Actue MeV Infection: Participants have acute MeV infection.
  Interventions: Biological: Verorab
- Group 2 - No Actue MeV Infection: Participants do not have acute MeV infection.
  Interventions: Biological: Verorab

INTERVENTIONS:
Biological: Verorab — Participants in each group will receive rabies vaccination (standard 3-dose series given as PrEP), with the first dose randomized to either Week 8 or Week 47 after enrollment.

SUMMARY:
The goal of this observational study is to investigate the effects of measles virus (MeV) infection on pre-existing immunity, vaccine response, and susceptibility to subsequent illness in children aged 1-15 either with or without acute MeV infection.

DETAILED DESCRIPTION:
This is a prospective, observational, longitudinal study to be conducted in West Africa. Eligible children will be enrolled into 1 of 2 arms: acute MeV infection (cases) or no acute MeV infection (controls) as assessed using upper respiratory specimens and blood samples. Blood samples will be collected at screening/enrollment (Day 0) and follow-up visits on Day 14, Week 13, and Week 52, and tested for humoral and cellular immune responses to endemic pathogens to determine changes in antibody diversity and antibody secreting cells (ASCs). All children in each arm will receive rabies vaccination (standard 3-dose series given as pre-exposure prophylaxis [PrEP]), with the first dose randomized to either Week 8 or Week 47 after enrollment. Biological samples will be collected after vaccination to assess if the immune stimulus (rabies vaccine) response differs: 1) between children with and without MeV infection, and 2) based on the timing of the receipt of the rabies vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1 to 15 years.
* Ability of the participant's legal or culturally acceptable representative to provide informed consent.
* Ability to give assent, as appropriate.
* Stated willingness of parent/guardian and participant as appropriate, to comply with all study procedures.
* Willingness to receive rabies vaccine.
* Meet the criteria for assignment to Group 1 or Group 2, as follows:
* Group 1, cases (acute MeV infection):
* Clinical signs and symptoms suggestive of acute MeV infection (Koplik spots or skin rash) AND
* Laboratory confirmed measles:
* Upper respiratory specimen (swab) PCR for measles positive, OR
* Serum IgM for measles positive.
* Group 2, controls (no acute MeV infection):
* No clinical signs and symptoms suggestive of acute MeV infection (Koplik spots or skin rash) AND
* Upper respiratory specimen (swab) PCR negative for MeV AND
* Serum measles IgM negative AND
* Serum measles IgG positive and previously vaccinated for measles (2nd dose will be offered if appropriate). If serum measles IgG is negative, participant must be willing to be vaccinated regardless of prior measles vaccine history to meet this criterion.

Exclusion Criteria:

* HIV infection or any other immunosuppressive condition or medications.
* Pregnant or lactating.
* History of prior measles or immunologic evidence of prior measles in the absence of prior measles vaccination.
* Severe anemia, defined as hemoglobin less than 8 g/dL.
* Any acute or chronic condition which, in the opinion of the investigator, constitutes a contraindication to participation in this study.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Specific study sites within each country will be in areas experiencing measles outbreaks.
Sampling Method: Non-Probability Sample
Enrollment: 256 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in pre-existing immunity | Week 13 after baseline
  Mean change in a panel of antibody levels over 13 weeks as measured by multiplex serological methods and targeted ELISAs for confirmation.
Effect of MeV infection on immune response to a controlled immune stimulus (rabies vaccination) | 14 days after last PrEP regimen vaccination
  Proportion of subjects with rabies virus neutralizing antibodies (RVNA) titer ≥ 0.5 IU/mL as measured by rapid fluorescent focus inhibition test
Effect of MeV infection on immune response to a controlled immune stimulus | 5-6 weeks after the first rabies vaccine dose
  Proportion of subjects with an RVNA titer ≥ lower limit of quantification
Effect of MeV infection on immune response to a controlled immune stimulus | 5-6 weeks after the first rabies vaccine dose
  Geometric mean RVNA titer

SECONDARY OUTCOMES:
Change in healthcare system encounters | 1 year following enrollment
  Mean number of non-study sick visit healthcare system encounters during the 1-year follow-up.
Change in pre-existing immunity | Week 52 after baseline
  Mean change in a panel of antibody levels over 52 weeks as measured by multiplex serological methods and targeted ELISAs for confirmation.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Hunsberger, Ph.D., Study Director — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- Partnership of Clinical Research in Guinea, Partenariat Pour La Recherche Clinique en Guinée (PREGUI), Conakry, Guinea
- University Clinical Research Center (UCRC) University of Sciences, Techniques and Technologies of Bamako, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tchos KF, Ridzon R, Haidara MC, Dabitao D, Akpa E, Camara D, Vallee D, Coulibaly M, Camara S, Aboulhab J, Diakite M, Diarra B, Diarra S, Dicko I, Francis A, Kolie CF, Koropogui M, Lim C, Samake S, Hunsberger S, Sidibe M, Chen RY, Konate I, Doumbia S, Beavogui AH, Shaw-Saliba K. Investigating immune amnesia after measles virus infection in two West African countries: A study protocol. PLoS One. 2025 Jun 26;20(6):e0314828. doi: 10.1371/journal.pone.0314828. eCollection 2025. PMID 40569945